CLINICAL TRIAL: NCT01589055
Title: IV Nicotine Induced Changes in Hormone Function, Mood States and Behavior
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects were ever enrolled; study not initiated
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Scott Lukas, Director, Alcohol and Drug Abuse Research Center & Professor of Psychology (Neuroscience), Harvard Medical School, Mclean Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2005-p-001057
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Last update posted 2024-01-17 (Actual); Status verified 2013-03

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Male Smokers (Active Comparator)
  Interventions: Drug: Intravenous Nicotine
- Female Smokers (Mid-Luteal Phase; cycle days 18-22) (Active Comparator)
  Interventions: Drug: Intravenous Nicotine
- Female Smokers (Early Follicular Phase; cycle days 4-8) (Active Comparator)
  Interventions: Drug: Intravenous Nicotine

INTERVENTIONS:
Drug: Intravenous Nicotine — Subjects will be given an intravenous challenge dose of nicotine or placebo in a constant volume of 1 ml on any study day. The nicotine solution (1.0 mg/70kg or 1.5 mg/70kg or 2.0 mg/70kg) will be administered over 1 min. This rate of drug delivery (1 ml over 1 min) has been safe in our IRB approved studies of nicotine. Most investigators have administered nicotine over 10 sec without any adverse reactions. We concur with the IRB recommendation that the lower doses (1.0 mg/70kg and 1.5 mg/70kg;) should be administered first and the higher dose (2.0 mg/70kg) will be administered last.
  Other Names: IV Nicotine

SUMMARY:
Clinical studies are proposed to analyze the interactions between nicotine, alterations in endocrine hormones, mood and cardiovascular measures. The studies are designed to examine the contribution of gender and menstrual cycle phase. It is hypothesized that analysis of nicotine's rapid hormonal, cardiovascular and subjective effects will be important for developing novel biologic approaches to treatment for nicotine abuse and dependence as well as advancing understanding of the neurobiology of nicotine reinforcement.

DETAILED DESCRIPTION:
These clinical studies are designed to examine the acute effects of intravenous nicotine on anterior pituitary (ACTH, LH) and adrenal hormones (DHEA and cortisol). We also plan to study norepinephrine (NE) and epinephrine (E), because nicotine stimulates rapid release of NE and E in preclinical and clinical studies. The studies will examine the acute effects of intravenous nicotine on the gonadal steroid hormones and the reciprocal feedback regulation by LH. The temporal covariance of hormonal changes with serum nicotine levels and nicotine-induced changes in subjective states and cardiovascular measures will be measured. The covariance between nicotine-induced changes in endocrine, subjective and cardiovascular effects and the temporal concordance with increases in serum nicotine and cotinine levels will be determined. Gender and menstrual cycle phase influences on the effects of nicotine on HPA and HPG hormones and subjective effects will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 40 who currently smoke at least 15 cigarettes every day, and who fulfill DSM-IV diagnostic criteria for nicotine dependence (305.10) will be eligible for participation.
* No evidence of clinically significant disease based upon complete medical history and physical examination by Dr. Arthur Siegel (Chief of Internal Medicine, McLean Hospital).
* Absence of DSM-IV Axis I Disorders other than nicotine dependence (305.10) as measured by the Structured Clinical Interview (SCID).
* Routine laboratory blood tests including complete blood count, electrolytes, BUN and creatinine, liver function test, hepatitis panel and urinalysis will be performed. Laboratory parameters must be within the normal range. HBsAg must be negative but subjects who have hepatitis serology consistent with previous exposure to Hepatitis A, Hepatitis B, or Hepatitis C, but who do not have clinical and biochemical evidence of acute infection, will be acceptable.
* Hematocrit levels ≥ 39% for males and ≥ 35% for females.
* Serum pregnancy test (hCG beta subunit) results must be negative within 24 hrs of the study day.
* Normal ECG.
* Subjects must be able to read and understand instructions, as well as provide a valid informed consent.

Exclusion Criteria:

* Women and men with any lifetime DSM-IV Axis I disorder other than nicotine abuse or dependence will be excluded.
* Women who are pregnant will be excluded.
* Women who use hormonal contraceptive medications will not be accepted for participation because this would confound the hormonal measures.
* Men and women with clinically significant medical disorders will be excluded.
* Obese and underweight subjects will be excluded. A mean Body Mass Index (ratio of weight (W) to height (H) squared; W/H2=kg/m2) will be calculated. Women with a mean Body Mass Index (BMI) of between 18.0-27.0 and men with a BMI between 21.4-29.0 will be accepted.
* Treatment seeking subjects will not be selected but will be referred to local smoking cessation programs.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2005-04; Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
Effects of nicotine on hormones and mood states | From baseline to study completion (approximately 4 months for males and 8 months for females)
  We are examining the effects of IV nicotine on serum nicotine levels, serum/plasma hormone levels and nicotine-induced changes in subjective statues, as measured by a visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy K M, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- Alcohol and Drug Abuse Research Center at McLean Hospital, Belmont, Massachusetts, United States